CLINICAL TRIAL: NCT03830541
Title: A Pattern of Oral Health Care Delivery for Persons With Autism Spectrum Disorder
Brief Title: Oral Health Care in Autism Spectrum Disorder
Acronym: CREASED
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Novi Sad (Other)
Responsible Party: Principal Investigator, Bojan Petrovic, Principal Investigator, University of Novi Sad
Other Study IDs: 01789/2019
Record Dates: First submitted 2019-02-02; First posted 2019-02-05 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-02

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: oral health; dental care; general anaesthesia; tooth loss
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Tooth Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Oral care delivery analysis in participants with ASD — The analysis of oral health status, tooth loss, oral rehabilitation, characteristics of routine dental treatment and treatment in general anaesthesia in persons with ASD

SUMMARY:
Persons with autism spectrum disorder (ASD) are characterized by impairments in social interactions, speech and communication, restricted patterns of behaviour, and unusual sensory sensitivities. There are not many studies available reporting oral health status, dental care needs and oral health care protocol for persons with an ASD.

DETAILED DESCRIPTION:
Despite the fact that there appears to be no known ASD specific dental and oral manifestations, there are consistent reports that persons with ASD exhibit significantly poorer oral health epidemiological profile when compared to their neurotypical counterparts. In addition to that, it has been reported that persons with ASD to substantial extent have a special health care needs and are almost twice as likely to have unmet oral health care needs as their typically developing peers regardless socioeconomic and cultural background. All these oral health related problems might arise because of ASD related challenging behaviors such as communication limitations, personal neglect, self-injurious behaviors, dietary habits, effects of medications, resistance to receiving dental care, hyposensitivity to pain, and possible avoidance of social contact. Frequently overlooked but very important reason is the lack of oral care providers who are willing to serve this population. As a results, oral health problems and unmet oral health needs transfer from childhood to adult period in persons with ASD.The broad, long-term objective of the investigator's proposed research is to describe the oral health status, oral health related behaviors, oral care delivery pattern, limitations of routine dental treatment and requirements for use general anaesthesia for oral health care of patients with ASD. Oral health status, pattern of oral health care delivery, dental treatment needs met in routine dental treatment and general anaesthesia will be analysed retrospectively on 52 participants with diagnosed ASD who were treated and monitored at the Paediatric Dentistry Department, Dental Clinic of Vojvodina, Faculty of Medicine, University of Novi Sad during 5 years (2013-2018) observation period. Conditions assessed will include, dental caries, missed teeth, filled teeth (DMFT index), restorations, bruxism, delayed eruption/missing teeth, oral infection, injuries, general health status, dental treatment acceptance (Frankle scale), dental treatment attendance, routine dental treatment and general anaesthesia dental treatment assessment.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Diagnosis of a autism spectrum disorder not confirmed by a physician

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with ASD treated at the Dental Clinic of Vojvodina during 5 years observation period
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2019-03-20 (Estimated); Primary Completion 2019-07-20 (Estimated); Study Completion 2019-12-20 (Estimated)

PRIMARY OUTCOMES:
Oral Health Status as measured by number of subjects with missing teeth | 3 months
  The number of missing teeth (T) is quantified using the D (decayed) component of the DMFT Index. The DMFT Index quantifies the dental caries experience by the number of decayed (D), missing (M), and filled (F) teeth (T). The number of subjects presenting with missing teeth will be reported.
Oral Health Status as measured by untreated dental decay | 6months
  Untreated dental decay will be determined by either the presence of coronal caries quantified by using the D (decayed teeth) component of the DMF (decayed, missed, filled) Index. The DMF Index quantifies the dental caries experience by the number of decayed (D), missing (M), and filled (F) teeth. The higher proportion of D in DMFT score suggest higher caries activity and poorer epidemiological profile
Oral health care delivery analysis | 3 months
  Reporting the mean numbers of regular dental treatment visits and general anesthesia treatment in various subgroups of participants

SECONDARY OUTCOMES:
Tooth loss in institutionalised participants | 3 months
  Comparison of proportions of permanent teeth extractions as calculated as T fraction in DMFT index between institutionalised and non institutionalised participants
Tooth loss in general anaesthesia | 6 months
  Comparison of proportions of permanent teeth extractions as calculated as T fraction in DMFT index between participants treated solely in general anaesthesia and participants exclusively treated during routine dental treatment

IPD SHARING:
Plan to Share IPD: No